CLINICAL TRIAL: NCT05799131
Title: QBX (5F/6F) Peripheral Balloon Expandable Stent System for the Treatment of Peripheral Artery Disease (PAD): Assessing Safety and Clinical Performance up to 12-months Follow-up
Brief Title: Safety and Efficacy of the QBX Peripheral Balloon Expandable Stent System in Peripheral Artery Disease (PAD)
Acronym: QBX-RADAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: QualiMed Innovative Medizinprodukte GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: QBX-RADAR
Record Dates: First submitted 2023-03-06; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QBX (5F/6F) Peripheral Balloon Expandable Stent System
  Interventions: Device: QBX (5F/6F) Peripheral Balloon Expandable Stent System

INTERVENTIONS:
Device: QBX (5F/6F) Peripheral Balloon Expandable Stent System — The QBX Stent System is a flexible, balloon expandable stent, made of a cobalt chromium alloy manufactured by QualiMed Innovative Medizinprodukte GmbH. The design is suitable for peripheral vessel diameters from 5 to 10 mm.
  The QBX Stent System is available as 6F and 5F variations where the 6F system is mounted on an 0.035" over-the-wire delivery system, and the 5F is mounted on an 0.018" over-the-wire delivery system. Both are available in a full range of diameters and lengths.

SUMMARY:
This study aims to evaluate the safety and performance of the QBX stent system in the treatment of PAD by reporting of peri- and postoperative complications, including major adverse vascular events (MAVE), Vascular Access Site Complications (VASCs) and bleeding at puncture site, and by evaluating the prevalence of Target Vessel Revascularization (TVR), amputations, procedural success, device performance, reduction in percentage diameter stenosis post-procedure compared to pre-procedure, artery patency, return to normal activity, Rutherford and Fontaine classification, quality of life (QoL), Ankle Brachial Index (ABI), and hospital- and patient-related costs in a prospectively maintained database.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for implantation of a peripheral balloon-expandable stent.
* Target lesion is an occlusion or diameter stenosis is ≥50% by visual estimate.
* Target lesion is a de novo or restenotic lesion.
* Target lesion is located in the external iliac artery (EIA), internal iliac artery (IIA), common iliac artery (CIA), superficial femoral artery (SFA) and/or deep femoral artery (DFA). Bilateral treatment of the target lesions is allowed. There are no restrictions on the number of target lesions treated with QBX or the number of stents used. Kissing stents and overlapping stents are allowed to treat the target lesions.
* Patient suffers from mild to intermittent claudication (Rutherford 1-3) or critical limb ischemia (Rutherford 4-5).
* Patients with TASC A, B, C and D lesions.
* Patient ≥ 18 years of age at study entry.
* Patient and investigator signed and dated the informed consent form prior to the index-procedure.

Exclusion Criteria:

* Age < 18 y.
* Pregnant women, women who are currently breastfeeding, women of childbearing potential who are not using an effective method of contraception, or women planning to become pregnant during the course of the study.
* Patients with Rutherford 0 and 6.
* Patient received a different stent device than the study device for the target lesion.
* Target lesion cannot be crossed with a guidewire (e.g. heavily calcified or excessively tortuous target lesion).
* Reference vessel diameter is not suitable for the available stent design.
* Target lesion was previously treated with a stent.
* Target lesion is in a prosthetic vascular bypass graft or within 1 cm of a graft anastomosis.
* Presence of significant stenosis (≥50%) or occlusion of inflow tract not successfully treated before or during the index-procedure (success is measured as < 30% residual stenosis and absence of distal embolization).
* Outflow: In case of treatment of iliac arteries: Inadequate distal runoff with > 50% stenosis of either the common femoral artery or both the superficial and deep femoral arteries. In case of treatment of the SFA: Absence of at least one patent runoff vessel with ≤ 50% stenosis throughout its course (i.e., confirmed in-line patency to the level of the foot). Outflow can be treated before or during the index-procedure (success is measured as < 30% residual stenosis and absence of distal embolization).
* Presence of active inflammation at the planned access site.
* Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index-procedure.
* Patients in severe renal failure (estimated Glomerular filtration rate (eGFR) < 25 mL/min/1.73m). Lab results are maximum 30 days old.
* Patient has a persistent acute intraluminal thrombus of the target lesion.
* Target lesion is in an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion.
* Patient has an abdominal aortic aneurysm contiguous with an iliac artery target lesion.
* Patient suffers from acute limb ischemia defined as any sudden decrease in limb perfusion causing a potential threat to limb viability.
* Contraindication for anti-coagulation therapy (coagulopathy, etc.).
* Patient has a known intolerance to contrast agents. If hypersensitivity to contrast agents in patients with prior reactions could be improved by premedication and changing the contrast agent, the patient can be included in the study.
* Patients has a known hypersensitivity to the stent material (L605).
* Patient has a life expectancy of <12 months.
* Patient has a planned surgical intervention/procedure, interfering with the study (results), within 30 days of the study procedure.
* Patient is considered to be hemodynamically unstable at onset of index-procedure.
* Patient is currently participating in a confounding study.
* Patient is unable to comply with the protocol or proposed follow-up visits.
* Patient is unable / unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PAD which are indicated to receive treatment with the QBX balloon-expandable stent and 5/6-French system through a femoral access with the aim to improve the vessel lumen diameter of target lesions (de novo and re-stenoses) in native peripheral arteries, e.g. external iliac artery (EIA), internal iliac artery (IIA), common iliac artery (CIA), superficial femoral artery (SFA) and deep femoral artery (DFA).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the cumulative rate of MAVE. | 12-months follow-up
  MAVE is defined as:
  1. Device- or procedure-related death;
  2. Target Lesion Revascularization (TLR) at 12 months, defined as a repeated procedure (endovascular or open surgery) due to a problem arising from the lesion (+1 cm proximally and distally to include edge phenomena) initially treated;
  3. Device-related distal embolization that required hospitalization and/or subsequent intervention.

SECONDARY OUTCOMES:
Rate of subjects with Vascular Access Site Complications (VASCs) within the first 24h after the index-procedure | 24 hours
  VASCs are defined as:
  * Hematoma/bleeding requiring transfusion
  * Arterial/venous occlusion/thrombosis
  * Severe vasospasm
  * Intimal injury/dissection
  * Pseudoaneurysm
  * Arteriovenous fistula
  * Vascular perforation or rupture
  * Arterial embolization distal to treatment site
  * Neuropathy
  * Retroperitoneal hematoma
Intra-operative complication rate. | Index-procedure
Post-operative complication rate. | 12-months follow-up
Intra-operative absence of bleeding at puncture site. | Index-procedure
Re-occlusion rate. | 12-months follow-up
  Re-occlusion is defined as complete occlusion of the target lesion initially treated.
Target Vessel Revascularization (TVR) rate. | 12-months follow-up
  TVR is defined as a procedure (endovascular or open surgical) due to a problem arising in the target vessel remote from the target lesion(s) initially treated.
Amputation rate | 12-months follow-up
  Minor (below the ankle) and major (above the ankle) amputation rate at 12 months will be assessed. Major amputation rates must be reported as below-the-knee and above-the-knee amputations.
Procedural success. | Index-procedure
  Procedural success is defined as a combination of technical success, device success and absence of procedural complications.
Technical success | Index-procedure
  Technical success is defined as successful vascular access and completion of the endovascular procedure and immediate morphological success with less than 30% residual diameter reduction of the treated lesion on completion angiography.
Device success. | Index-procedure
  Device success is defined as exact deployment of the device according to the instructions for use.
Device performance. | Index-procedure
  Scored using the following components and a dedicated Scoring System (1: Very good, 2: Good, 3: Sufficient, Poor: 4):
  * Insertion through introducer sheath
  * Tracking to target site over guidewire
  * Crossability through of the lesion
  * Catheter pushability
  * Catheter shaft kink resistance
  * Stent radiopacity
  * Inflation time to Nominal diameter
  * Deflation time
  * Stent apposition
  * General usability of the QBX device
Reduction in percentage diameter stenosis post-procedure compared to pre-procedure. | Index-procedure
  Assessed via CT angio.
Artery patency. | 1-month follow-up
  A duplex ultrasound will be performed to evaluate artery patency. If reliable duplex ultrasound assessment of artery patency is not possible, ABI is a good indication of patency. If ABI is abnormal and the patient is experiencing symptoms, a CT angio or other imaging module might be performed according to standard of care.
Artery patency. | 6-months follow-up
  A duplex ultrasound will be performed to evaluate artery patency. If reliable duplex ultrasound assessment of artery patency is not possible, ABI is a good indication of patency. If ABI is abnormal and the patient is experiencing symptoms, a CT angio or other imaging module might be performed according to standard of care.
Artery patency. | 12-months follow-up
  A duplex ultrasound will be performed to evaluate artery patency. If reliable duplex ultrasound assessment of artery patency is not possible, ABI is a good indication of patency. If ABI is abnormal and the patient is experiencing symptoms, a CT angio or other imaging module might be performed according to standard of care.
Return to normal activity. | 1-month follow-up
  The number of days until return to normal activities will be assessed.
Distribution of Rutherford classes during follow-up as compared to baseline. | 1-month follow-up
  The percentage of patients with Rutherford classes 0 to 6 will be determined.
Distribution of Rutherford classes during follow-up as compared to baseline. | 6-months follow-up
  The percentage of patients with Rutherford classes 0 to 6 will be determined.
Distribution of Rutherford classes during follow-up as compared to baseline. | 12-months follow-up
  The percentage of patients with Rutherford classes 0 to 6 will be determined.
Distribution of Fontaine stages during follow-up as compared to baseline. | 1-month follow-up
  The percentage of patients with Fontaine stages I to IV will be determined.
Distribution of Fontaine stages during follow-up as compared to baseline. | 6-months follow-up
  The percentage of patients with Fontaine stages I to IV will be determined.
Distribution of Fontaine stages during follow-up as compared to baseline. | 12-months follow-up
  The percentage of patients with Fontaine stages I to IV will be determined.
Primary sustained clinical improvement at 12 months. | 12-months follow-up
  Primary sustained clinical improvement is defined as sustained upward shift of at least one category on the Rutherford/Fontaine classification without the need for repeated TLR in surviving patients.
Secondary sustained clinical improvement at 12 months. | 12-months follow-up
  Secondary sustained clinical improvement is defined as sustained upward shift of at least one category on the Rutherford/Fontaine classification including the need for repeated TLR in surviving patients.
Improvement in disease-related health status, functioning and quality of life at follow-up as compared to baseline. | 1-month follow-up
  This is scored by the Walking Impairment Questionnaire and EQ-5D questionnaire.
Improvement in disease-related health status, functioning and quality of life at follow-up as compared to baseline. | 6-months follow-up
  This is scored by the Walking Impairment Questionnaire and EQ-5D questionnaire.
Improvement in disease-related health status, functioning and quality of life at follow-up as compared to baseline. | 12-months follow-up
  This is scored by the Walking Impairment Questionnaire and EQ-5D questionnaire.
Ankle Brachial Index (ABI) during follow-up as compared to baseline. | 1-month follow-up
Ankle Brachial Index (ABI) during follow-up as compared to baseline. | 6-months follow-up
Ankle Brachial Index (ABI) during follow-up as compared to baseline. | 12-months follow-up
Occurrence of prolonged hospitalization compared to local standard of care (SOC). | Immediately after the procedure
  When the patient leaves the hospital after the procedure.
Time taken off from work for the procedure | 1-month follow-up
  Consists of:
  * Initial sick leave after the surgery
  * Additional sick leave
  * Leave taken by friends/relatives for patient care

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - Ziekenhuis Oost-Limburg Genk, Genk, Limburg
  - Jessa Ziekenhuis, Hasselt, Limburg
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - HIS IZZ, Brussels